CLINICAL TRIAL: NCT06178692
Title: Validation Study of a Serum-miRNA Signature, Associated With IDH1 Stuatus, as Non-invasive Diagnostic and Prognostic Biomarkers in Glioma Patients
Brief Title: Validation Study of a Serum-miRNA Signature in Glioma Patients.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Azienda Ospedaliero Universitaria di Sassari (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); University of Roma La Sapienza (Other); Plymouth State University (Other)
Responsible Party: Sponsor
Other Study IDs: RS1337/20
Record Dates: First submitted 2023-03-28; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Biomarker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples: two test tubes (6ml each) with activator of peripheral blood coagulation at diagnosis, at discharge after surgery (4-6 days after surgery) and/or at the first post-surgery check-up. From the serum obtained from blood samples will subsequently be extracted the RNA and the expression level of the miRNAs will be analyzed in individual samples by digital PCR.
  * Tissue samples: where possible, biopsy tissue taken for diagnostic purposes and fixed in formalin and embedded in paraffin (FFPE) will be analyzed for the expression of miRNAs of interest by Real-Time PCR.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: IDH1 mutated
  Interventions: Diagnostic Test: Validation of miRNA-serum signatures associated with IDH1 status
- Arm 2: IDH1 wt
  Interventions: Diagnostic Test: Validation of miRNA-serum signatures associated with IDH1 status

INTERVENTIONS:
Diagnostic Test: Validation of miRNA-serum signatures associated with IDH1 status — Validation of miRNA-serum signatures associated with IDH1 status and prognosis, as reliable, specific and sensitive circulating diagnostic biomarkers also useful to improve prognostic stratification of patients.

SUMMARY:
Prospective, multicenter, noninterventional, nonprofit study of a cohort of patients with glioma, aimed at validating miRNA-serum signatures associated with IDH1 status and prognosis, as reliable, specific and sensitive circulating diagnostic biomarkers also useful for improve prognostic stratification of patients. The study will be conducted on serum samples at diagnosis, at 4-6 days postoperatively and/or at the first post-surgery follow-up, in a new cohort of glioma patients and representative of different IDH1 mutational statuses. Furthermore, because comparison of miRNA expression profiles in serum and tissue may provide further evidence to support the use of serum miRNAs as reliable biomarkers reliable, their expression will also be analyzed, where possible, in tissue biopsies from the same patient and compared with the expression profiles of serum miRNAs.

DETAILED DESCRIPTION:
Scientific data suggest that a serum signature of miRNA could be a promising noninvasive diagnostic and prognostic tool for stratify, by liquid biopsy, patients with glioma according to IDH1 status. It has the primary objective of validating, through non-invasive methods, a signature of Serum miRNAs as reliable, specific and sensitive diagnostic and/or prognostic biomarkers for patients affected by glioma which can also help integrate the molecular analyzes performed on biopsies tissue. The ultimate goal is therefore to validate specific biomarkers for a "medicine" approach personalized" for glioma patients, with potential clinical benefits resulting from improved patient management and identification of the best possible therapy for specific subgroups biological data of patients. Blood samples from cancer patients will be used brain with different IDH1 status and of different grade, recruited from the centers participating in the study.

Where possible, tissue samples coming, according to clinical practice, from biopsy will be used to the diagnosis of the same patient.

For the analyzes foreseen by the study it will be necessary to take two test tubes (6ml each) with activator of peripheral blood coagulation at diagnosis, at discharge after surgery (4-6 days after surgery) and/or at the first post-surgery check-up. From the serum obtained from blood samples will subsequently be extracted the RNA and the expression level of the miRNAs will be analyzed in individual samples by digital PCR.

The method of collection of peripheral blood samples at diagnosis, discharge and/or following the first post-surgery check-up it will be kept uniform throughout study, to minimize preanalytical variables. Any hemolyzed samples will be identified, and excluded from the study, through spectrophotometric analysis and/or by analyzing the level of expression of miR-451, abundant in erythrocytes, and miR-23a, not affected by hemolysis.

Where possible, biopsy tissue taken for diagnostic purposes and fixed in formalin and embedded in paraffin (FFPE) will be analyzed for the expression of miRNAs of interest by Real-Time PCR.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of glioma;
* age≥18 years;
* No other primary tumor;
* No metastatic disease
* Informed consent on treatment and molecular analysis

Exclusion Criteria:

* Histological diagnosis of non-glial tumor;
* age< 18;
* patients with concomitant other solid tumors
* metastatic disease; HIV seropositivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective, multicenter, noninterventional, nonprofit study of a cohort of patients with glioma, aimed at validating miRNA-serum signatures associated with IDH1 status and prognosis, as reliable, specific and sensitive circulating diagnostic biomarkers also useful for improve prognostic stratification of patients.
  The study will be conducted on serum samples at diagnosis, at 4-6 days postoperatively and/or at the first post-surgery follow-up, in a new cohort of glioma patients and representative of different IDH1 mutational statuses.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Identification of specific forms of circulating microRNAs invasive brain tumors | Enlistment period: 6-12 months Total duration of the study: 18-24 months
  Identification of specific circulating microRNA signatures as non-diagnostic biomarkers invasive brain tumors.
  The variables of interest will be summarized by descriptive statistics. ROC curve analysis will be used to evaluate the diagnostic accuracy of miRNAs to be validated. Survival analysis (Overall Survival=OS and Progression Free Survival=PFS) will be conducted through the use of the Kaplan-Meier model and risk regression models Cox proportionals. The log-rank test will be used to test for any differences between groups. The Hazard Risk (HR) and related 95% confidence intervals (95%CI) will be estimated for each variable using univariate and multivariate Cox models. A p value <0.05 will be considered statistically significant. All analyzes will be conducted with SPSS v.21.0 software.

SECONDARY OUTCOMES:
Transfer of information in the clinical setting for diagnosis | Enlistment period: 6-12 months Total duration of the study: 18-24 months
  Transfer of this information into the clinical setting for diagnosis, prognosis and purposes therapeutic.
  The variables of interest will be summarized by descriptive statistics. ROC curve analysis will be used to evaluate the diagnostic accuracy of miRNAs to be validated. Survival analysis (Overall Survival=OS and Progression Free Survival=PFS) will be conducted through the use of the Kaplan-Meier model and risk regression models Cox proportionals. The log-rank test will be used to test for any differences between groups. The Hazard Risk (HR) and related 95% confidence intervals (95%CI) will be estimated for each variable using univariate and multivariate Cox models. A p value <0.05 will be considered statistically significant. All analyzes will be conducted with SPSS v.21.0 software.
Implementation of clinical trials leveraging know-how. | Enlistment period: 6-12 months Total duration of the study: 18-24 months
  Implementation and interpretation of clinical trials using specific know-how generated by the collaborative effort of study participants.
  The variables of interest will be summarized by descriptive statistics. ROC curve analysis will be used to evaluate the diagnostic accuracy of miRNAs to be validated. Survival analysis (Overall Survival=OS and Progression Free Survival=PFS) will be conducted through the use of the Kaplan-Meier model and risk regression models Cox proportionals. The log-rank test will be used to test for any differences between groups. The Hazard Risk (HR) and related 95% confidence intervals (95%CI) will be estimated for each variable using univariate and multivariate Cox models. A p value <0.05 will be considered statistically significant. All analyzes will be conducted with SPSS v.21.0 software.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Giulia Rizzo, Doctor, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided